CLINICAL TRIAL: NCT04190342
Title: Effects of a Traditional Chinese Exercise Program- Tai Chi on Symptom Cluster of Fatigue-sleep Disturbance-depression in Female Breast Cancer Patients: a Preliminary Randomized Controlled Trial
Brief Title: Effects of a Traditional Chinese Exercise Program on Symptom Cluster in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Darwin University (Other)
Collaborators: The Affiliated Hospital Of Southwest Medical University (Other); The Affiliated Hospital of Putian University (Other)
Responsible Party: Principal Investigator, Jing-Yu Tan, BNSc, MMed, PhD, Professor in Nursing, Charles Darwin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H19094
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Breast Neoplasm Female; Symptom Cluster; Tai ji
Keywords: tai chi; breast cancer; symptom cluster; fatigue; sleep disturbance; depression
MeSH Terms: conditions — Syndrome; Breast Neoplasms; Fatigue; Parasomnias; Depression | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): standard care (intervention provided after the completion of the trial)
  Interventions: Other: control group
- tai chi group (Experimental): Tai chi intervention + standard care
  Interventions: Behavioral: tai chi group

INTERVENTIONS:
Other: control group — A booklet on the self-management of cancer symptoms. After the pilot RCT is completed, if the participants allocated to the control group are interested in practising tai chi, the intervention will be provided
  Arms: control group
Behavioral: tai chi group — Around 60 minutes practising easy tai chi movements/postures twice per week
  Arms: tai chi group

SUMMARY:
The Medical Research Council Framework for Developing and Evaluating Complex Interventions (MRC Framework) will be utilized to develop and evaluate an evidence-based tai chi intervention for managing the symptom cluster of fatigue-sleep disturbance-depression in breast cancer patients.

DETAILED DESCRIPTION:
The fatigue-sleep disturbance-depression symptom cluster (FSDSC) is regarded as one of the most common symptom clusters among breast cancer (BC) patients. Considering the fact that no specific medications can be recommended to relieve symptom clusters, numerous non-pharmacological interventions have therefore been performed with medication as a combination intervention for the treatment of symptom clusters in cancer patients. Among these interventions, tai chi could be an optimal option for relieving the FSDSC. The overall aims are to develop an evidence-based traditional Chinese exercise (TCE) tai chi protocol, test the feasibility of the protocol, and preliminarily examine the effectiveness of tai chi on the FSDSC and quality of life (QoL) through a pilot randomized controlled trial (RCT). The MRC Framework will be used to develop and evaluate an evidence-based intervention for BC patients. In phase one, an evidence-based TCE tai chi intervention protocol will be developed. An expert panel will then be invited to assess the content validity of the intervention protocol. Testing the feasibility of the tai chi intervention protocol, and preliminarily examining the effects of tai chi on the FSDSC will be conducted in phase two. After completion of the pilot RCT, semi-structured interviews will be conducted to assess the participants' experience of participating in the pilot trial and performing the tai chi exercise. The evidence-based tai chi intervention protocol for managing the FSDSC in breast cancer patients will be developed. The feasibility and effects of utilizing the tai chi intervention for BC patients will be explored. A future multicentre large-scale RCT to further evaluate the effects of tai chi on the FSDSC in the BC population will benefit from the study results of this doctoral research project.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 18 years old or above;
2. a confirmed diagnosis of non-metastatic stage I, II, or IIIa BC;
3. have experienced at least a moderate level of tiredness, sleep disturbance, and depressive mood, with a score of greater than 3 on a 10-point numeric rating scale, from "0 (no symptom)" to "10 (worst symptom)" for each symptom in the previous one month;
4. have recently commenced adjuvant chemotherapy; and
5. able to follow instructions in Mandarin, interested in participating in the study, and willing to sign an informed consent.

Exclusion Criteria:

1. Currently using psychostimulants, antidepressant medications, or hypnotics medications;
2. extremely weak or have mental illness and/or intellectual disability;
3. have been involved in other exercise programs > 30 minutes, three times weekly, for past 3 months;
4. have practised tai chi for the past six months; and
5. have scheduled elective surgery during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Time taken to recruit planned sample | From baseline (T1) to the completion of the 8-week intervention (T2)
  the time that was taken to recruit the planned sample size of participants
Referral rate | From baseline (T1) to the completion of the 8-week intervention (T2)
  The number of referrals made by clinicians in different departments and hospitals divided by all referrals
Recruitment rate | From baseline (T1) to the completion of the 8-week intervention (T2)
  The number of subjects who enrolled in the study divided by all subjects eligible for enrolment
Retention rate | From baseline (T1) to the completion of the 8-week intervention (T2)
  The number of subjects who completed the study divided by all subjects who enrolled in the study
Dropout rate | From baseline (T1) to the completion of the 8-week intervention (T2)
  The number of subjects who dropped out after randomization divided by all subjects who enrolled in the study
Reasons for dropping out | From baseline (T1) to the completion of the 8-week intervention (T2)
  Feedback from the dropout subjects to identify their reasons for dropping out
Feasibility of the questionnaires | Baseline (T1), immediately after completion of the 8-week intervention (T2), and four weeks after completion of the intervention (T3)
  The percentage of missing values for each item of the scales used, including the Brief Fatigue Inventory (BFI), the Pittsburgh Sleep Quality Index (PSQI), the Hospital Anxiety and Depression Scale (HADS), and the Functional Assessment of Cancer Therapy-Breast (FACT-B)
Adherence rates | Immediately after completion of the 8-week intervention (T2)
  The adherence rates will be measured by the number of tai chi sessions performed divided by the total possible tai chi sessions
Participant feedback | Immediately after completion of the 8-week intervention (T2)
  Participants' feedback on and satisfaction with the intervention using a self-designed feedback form
Adverse events associated with the intervention | Immediately after completion of the 8-week intervention (T2)
  In each tai chi session, the subjects in the intervention group will record whether they had any uncomfortable feelings
Number of patients completed the exercise log | Immediately after completion of the 8-week intervention (T2)
  The participants in the tai chi group will be required to keep a diary to monitor their tai chi exercise after each tai chi session

SECONDARY OUTCOMES:
Symptom cluster assessment: fatigue | Baseline Assessments (T1); Immediately after completion of the 8-week intervention (T2); 4-week Follow-up (T3)
  Fatigue will be measured by the Brief Fatigue Inventory (BFI). The Brief Fatigue Inventory includes nine items using a 0- to 10-point Likert scale, where 0 = "no fatigue" and 10 = "fatigue as bad as you can imagine" . The global BFI score, with a range between 0 and 90, is calculated as the mean of the nine items, and higher scores correspond to more severe fatigue
Symptom cluster assessment: sleep disturbance | Baseline Assessments (T1); Immediately after completion of the 8-week intervention (T2); 4-week Follow-up (T3)
  Sleep disturbance will be measured by the Pittsburgh Sleep Quality Index (PSQI). This 19-item questionnaire consists of seven components: subjective sleep quality (one item), sleep latency (two items), sleep duration (one item), habitual sleep efficiency (three items), sleep disturbance (nine items), use of sleeping medications (one item), and daytime dysfunction (two items). Each of the seven component scores are identified based on scoring algorithms, with each item using a 4-point Likert response scale, ranging from 0 to 3. A global (total) score is obtained from the sum of the seven component scores, with a possible range of 0 to 21 points. A higher score on the global (total) score indicates poorer sleep quality.
Symptom cluster assessment: depression | Baseline Assessments (T1); Immediately after completion of the 8-week intervention (T2); 4-week Follow-up (T3)
  depression will be measured by the Hospital Anxiety and Depression Scale (HADS). The HADS is a 14-item, self-report scale that includes two subscales, namely, the Anxiety subscale (HADS-A) and the depression subscale (HADS-D), which has seven items per subscale. The scale uses a 4-point Likert scale, ranging from 0 to 3. The sum of the ratings of 14 items yields a total score; the sum of the ratings of seven items in each subscale yields separate scores for anxiety and depression. The score ranges between 0 and 42 for the total score and between 0 and 21 for each subscale. Higher scores indicate greater severity of anxiety and depression.
Quality of life (QoL) assessment | Baseline Assessments (T1); Immediately after completion of the 8-week intervention (T2); 4-week Follow-up (T3)
  Quality of life assessment will be measured by the Functional Assessment of Cancer Therapy-Breast (FACT-B). The FACT-B is subdivided into four primary QoL domains, namely, Physical Well-Being (seven items), Social Well-Being (seven items), Emotional Well-Being (six items), and Functional Well-Being (seven items), and contains additional concerns for Beast Cancer (10 items) . The FACT-B has a 5-point Likert-type response scale, ranging from 0 to 4, where 0 = "not at all" and 4 = "very much". A summing-up of each FACT-B subscale creates the FACT-B total score, ranging from 0 to 148. Moreover, a higher FACT-B score indicates a better QoL status.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Yu (Benjamin) Tan, PhD, Principal Investigator — Charles Darwin University
Locations (2):
- China (2):
  - The Affiliated Hospital of Putian University, Putian, Fujian
  - The Affiliated Hospital Of Southwest Medical University, Luzhou, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yao LQ, Tan JB, Turner C, Wang T. Feasibility and potential effects of tai chi for the fatigue-sleep disturbance-depression symptom cluster in patients with breast cancer: protocol of a preliminary randomised controlled trial. BMJ Open. 2021 Aug 18;11(8):e048115. doi: 10.1136/bmjopen-2020-048115. PMID 34408044